CLINICAL TRIAL: NCT06688682
Title: Effect of PRP Joint Cavity Combined with Acupoint Injection on Osteoarthritis of Knee Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhengzhou Revo-Gene Technology Co., LTD (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RG2301
Record Dates: First submitted 2024-11-09; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Early Knee Osseous Arthrophlogosis
MeSH Terms: interventions — Acupuncture Points

STUDY DESIGN:
Intervention Model Description: 90 subjects were randomly divided into three groups, with 30 cases in each group. (1) HA group: The patients were given intraarticular injection of sodium hyaluronate injection, 2ml each time, and normal saline injection of 1ml at Xuehai point, Yanglingquan point and Wezhong point, once a week for 4 weeks. (2) PRP joint cavity injection group: PRP knee cavity injection was given, 3.5ml each time, and normal saline injection was given at Xuechai point, Yanglingquan point and Weizhong point 1ml, once a week for 4 weeks; (3) PRP joint cavity combined with acupoint injection group: PRP was given intraventricular injection of knee joint, each injection was 3.5ml, while PRP was given 1ml injection of Xuehai point, Yanglingquan point and Weizhong point, once a week for 4 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HA group (No Intervention): treated with intra-articular injection of hyaluronic acid solution, 2 ml per injection, and 1 ml of normal saline injection at Xuehai, Yanglingquan, and Weizhong acupoints at the same time, once a week for 4 weeks
- PRP joint injection group (Placebo Comparator): treated with intra-articular injection of PRP, 3.5 ml per injection, and 1 ml of normal saline injection at Xuehai, Yanglingquan, and Weizhong acupoints at the same time, once a week for 4 weeks
  Interventions: Other: PRP joint injection combined with acupoint injection
- PRP joint injection combined with acupoint injection group (Experimental): treated with intra-articular injection of PRP, 3.5 ml per injection, and 1 ml of PRP injection at Xuehai, Yanglingquan, and Weizhong acupoints at the same time, once a week for 4 weeks
  Interventions: Other: PRP joint injection combined with acupoint injection

INTERVENTIONS:
Other: PRP joint injection combined with acupoint injection — PRP acupoint injection
  Arms: PRP joint injection combined with acupoint injection group; PRP joint injection group

SUMMARY:
This study collected general data from 90 patients with KOA in the outpatients and ward of Henan Provincial People's Hospital from January 2023 to December 2023 to compare the long-term effects of intra-articular PRP combined with acupoint PRP, intra-articular PRP, and intra-articular HA on symptoms in patients with mild to moderate osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

1. The expected survival period is more than 3 months;
2. The clinical diagnosis was early knee osteoarthritis;
3. Capable of knee injections;
4. chronic joint pain or swelling (> 4 months);
5. It meets the diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of Osteoarthritis (2021 Edition) , and the X-ray evaluation results meet the Kellgren-Lawrence scale (K-L scale) level I to level III.

Exclusion Criteria:

1. age over 80 years old;
2. K-L classification is greater than Ⅲ grade;
3. Combined with rheumatoid arthritis, severe osteoporosis, tumor, gout, obvious joint deformity and other diseases;
4. Poor compliance, not according to the provisions of treatment;
5. Pregnant and lactating women;
6. Patients voluntarily withdrew from the study;
7. Patients were lost to follow-up due to various reasons during follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) score | Assessments will be conducted at weeks 1, 3, 6, and 12 after treatment.
  Visual Analog Scale (VAS) score ranging from 1 to 10, with lower scores indicating less pain intensity
Knee Society Score (KSS) | Assessments will be conducted at weeks 1, 3, 6, and 12 after treatment.
  Knee Society Score (KSS), which consists of five major items totaling 200 points. Higher scores indicate better knee joint function
Western Ontario and McMaster Universities Osteoarthritis Index | Assessments will be conducted at 1, 3, 6, and 12 months after treatment.
  The severity of knee osteoarthritis was measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score, consisting of 24 items with a total possible score of 240 points. Lower WOMAC scores indicate less severe knee osteoarthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- No.7, Wei Wu Road, Zhengzhou City, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No